CLINICAL TRIAL: NCT07217223
Title: Spaced Transcranial Direct Current Stimulation for Treatment-Resistant Depression: A Home-Based Feasibility and Safety Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jean-Philippe Miron, MD, PhD, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 812687; 812687 (Registry Identifier: Spaced Transcranial Direct Current Stimulation for Treatment-Resistant Depression: A Home-Based Feasibility and Safety)
Record Dates: First submitted 2025-09-30; First posted 2025-10-15 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-08

CONDITIONS: Treatment Resistant Depression (TRD); Major Depressive Disorder (MDD)
Keywords: Treatment; Treatment Resistant Depression; Major Depressive Disorder; MDD
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Spaced Transcranial Direct Current Stimulation Treatment (Experimental): tDCS, a non-invasive neuromodulation technique that applies low-intensity, direct electrical stimulation to the cortex via scalp electrodes, has been extensively researched as a potential treatment for MDD. tDCS enhances neuroplasticity, which is theorized to be responsible for its therapeutic effects and has been presented as a cost-effective solution for MDD. Preclinical evidence supports the potential advantage of spaced stimulation with tDCS to maximally engage neuroplasticity.
  tDCS sessions will be self-administered at home under the supervision of a trained clinical research coordinator.
  Each treatment day will consist of five tDCS sessions, each lasting 20 minutes, spaced by approximately 20-minute inter-session intervals, for a total of three hours per day.
  Other Names:
  * tDCS
  * Soterix Medical miniCT
  Interventions: Device: Spaced Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Spaced Transcranial Direct Current Stimulation (tDCS) — tDCS will be self-administered at home under the supervision of a trained clinical research coordinator using the Soterix Medical mini-CT device with remote monitoring via a secure videoconferencing platform (e.g., Microsoft Teams).The device is designed for safe, remote tDCS delivery. Participants will be treated using a stimulation at 2 mA, with a 30-second ramp-up and ramp-down phase.

SUMMARY:
The investigators propose a single-arm, open-label study to evaluate the effectiveness, safety, tolerability and feasibility of at-home transcranial direct current stimulation (tDCS) as a treatment for depression, particularly in cases where patients have not responded well to traditional therapies. Treatment will be delivered over a 2-week period with daily weekday treatments i.e., five tDCS sessions, each lasting 20 minutes, spaced by approximately 20-minute inter-session intervals, for a total of three hours a day. Participants will self-administer treatment at home under direct remote supervision. Pre- and post- treatment neurophysiological biomarkers sessions will also be carried out. The study aims to examine changes in mood, brain activity, and related clinical outcomes before, during, and after treatment, with the goal to provide more information that can be used for future studies.

PLEASE NOTE: THERE WILL BE 4 APPOINTMENTS THAT MUST OCCUR IN PERSON IN SAN DIEGO, CA.

ELIGIBILITY:
Inclusion Criteria:

1. People between the ages of 18 and 85 at the time of screening.
2. Currently diagnosed with Major Depressive Disorder (MDD) as measured by the MINI and a MADRS score of ≥ 20.
3. Safe for TMS as measures by the TMS Adult Safety Screening (TASS).
4. Medical records confirming a history of failing to achieve clinical response to an adequate antidepressant trial as defined an Antidepressant Treatment History Form (ATHF) score ≥ 3 or ) or shown intolerance to at least two inadequate trials (score 1 or 2), without psychiatric illness due to a general medical condition.
5. Stable internet connection and a device compatible with Microsoft Teams.

Exclusion Criteria:

1. History of psychotic or bipolar disorder or depression with psychotic features;
2. Significant borderline personality disorder;
3. Significant comorbid obsessive-compulsive or post-traumatic stress:
4. Current moderate or severe substance use disorder or demonstrating signs of acute substance withdrawal;
5. Clinically significant suicidality disorder;
6. Chronic depression (defined as of over 5 years duration);
7. Pregnancy or lactation, lack of adequate birth control in women of childbearing age;
8. History of significant neurologic disease, including dementia, Parkinson's or Huntington's disease, brain tumor, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma with persistent symptoms;
9. Unstable medical illness;
10. Contraindication to receiving tDCS (e.g., ferromagnetic implant, history of seizure, known brain lesion);
11. History of TMS (greater than 15 sessions) without a clinically meaningful response.; History of ketamine (greater than 4 sessions) without a clinically meaningful response;
12. Require a benzodiazepine with a dose > lorazepam 2 mg/day;
13. dermatological conditions contraindicating tDCS;
14. Non-correctable sensory impairments;
15. Inability to consent or participate as an outpatient

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-27 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility (Recruitment) | From baseline clinical assessment prior to treatment to 12 weeks after last treatment.
  Recruitment rate will be measured as the number of patients enrolled by the conclusion of the study, reported as a whole number.
Feasibility (Retention) | From baseline clinical assessment prior to treatment, to 12 weeks after last treatment.
  Retention rate will be measured as the percentage of enrolled patients who complete all study visits, reported as a percentage.
Feasibility (Adherence) | From baseline clinical assessment prior to treatment, to 12 weeks after last treatment.
  The proportion of completed sessions relative to the total prescribed sessions, expressed as a percentage.
Safety of at-home spaced tDCS | From baseline clinical assessment prior to treatment, to 12 weeks after last treatment.
  Safety will be measured by the number of serious adverse events (SAEs)
Tolerability to spaced tDCS | From baseline clinical assessment prior to treatment, to 12 weeks after last treatment.
  Tolerability will be measured by the number of adverse events (AEs).

SECONDARY OUTCOMES:
Changes from pre-treatment depressive symptomatology in post-treatment | From baseline clinical assessment prior to treatment, to 12 weeks after last treatment.
  Changes in depressive symptoms will be assessed using the Montgomery-Åsberg Depression Rating Scale (MADRS), which ranges from 0 to 60, with higher scores indicating more severe depression. A decrease in the MADRS score will be interpreted as an improvement in symptoms.
Biomarker Discovery: Short-Interval Intracortical Inhibition (SICI) via TMS-EMG | From baseline neurophysiological assessment prior to treatment, to during treatment, to 12 weeks after last treatment.
  TMS-EMG will be used to evaluate changes in SICI.
Biomarker Discovery: Intracortical Facilitation (ICF) via TMS-EMG | From baseline neurophysiological assessment prior to treatment, to during treatment, to 12 weeks after last treatment.
  TMS-EMG will be used to evaluate changes in intracortical facilitation
Biomarker Discovery: Cortical Silent Period (CSP) via Transcranial Magnetic Stimulation-Electromyography (TMS-EMG) | From baseline neurophysiological assessment prior to treatment, to during treatment, to 12 weeks after last treatment.
  TMS-EMG will be used to assess changes in the cortical silent period (CSP).
  Unit of Measurement: Duration (milliseconds).
Biomarker Discovery: TMS-Evoked Potential (TEP) Component Amplitudes via TMS-EEG | From baseline neurophysiological assessment prior to treatment, to during treatment, to 12 weeks after last treatment.
  TMS-EEG will be used to evaluate changes in TMS-evoked potential (TEP) component amplitudes.
  Unit of Measurement: Voltage (µV).
Biomarker Discovery: Resting-State Electroencephalography (rsEEG) | From baseline neurophysiological assessment prior to treatment, to during treatment, to 12 weeks after last treatment.
  rsEEG will be used to analyze changes in brain activity patterns at rest.
  Unit of Measurement: Frequency (Hz)
Biomarker Discovery: Resting-State Electroencephalography (rsEEG) | From baseline neurophysiological assessment prior to treatment, to during treatment, to 12 weeks after last treatment.
  rsEEG will be used to analyze changes in brain activity patterns at rest.
  Unit of Measurement: Amplitude (µV).

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Interventional Psychiatry, San Diego, California, United States

REFERENCES:
- [Background] Stagg CJ, Antal A, Nitsche MA. Physiology of Transcranial Direct Current Stimulation. J ECT. 2018 Sep;34(3):144-152. doi: 10.1097/YCT.0000000000000510. PMID 29877965
- [Background] Williams NR, Sudheimer KD, Bentzley BS, Pannu J, Stimpson KH, Duvio D, Cherian K, Hawkins J, Scherrer KH, Vyssoki B, DeSouza D, Raj KS, Keller J, Schatzberg AF. High-dose spaced theta-burst TMS as a rapid-acting antidepressant in highly refractory depression. Brain. 2018 Mar 1;141(3):e18. doi: 10.1093/brain/awx379. No abstract available. PMID 29415152
- [Background] Brunoni AR, Valiengo L, Baccaro A, Zanao TA, de Oliveira JF, Goulart A, Boggio PS, Lotufo PA, Bensenor IM, Fregni F. The sertraline vs. electrical current therapy for treating depression clinical study: results from a factorial, randomized, controlled trial. JAMA Psychiatry. 2013 Apr;70(4):383-91. doi: 10.1001/2013.jamapsychiatry.32. PMID 23389323
- [Background] Brunoni AR, Moffa AH, Sampaio-Junior B, Borrione L, Moreno ML, Fernandes RA, Veronezi BP, Nogueira BS, Aparicio LVM, Razza LB, Chamorro R, Tort LC, Fraguas R, Lotufo PA, Gattaz WF, Fregni F, Bensenor IM; ELECT-TDCS Investigators. Trial of Electrical Direct-Current Therapy versus Escitalopram for Depression. N Engl J Med. 2017 Jun 29;376(26):2523-2533. doi: 10.1056/NEJMoa1612999. PMID 28657871
- [Background] Fritsch B, Reis J, Martinowich K, Schambra HM, Ji Y, Cohen LG, Lu B. Direct current stimulation promotes BDNF-dependent synaptic plasticity: potential implications for motor learning. Neuron. 2010 Apr 29;66(2):198-204. doi: 10.1016/j.neuron.2010.03.035. PMID 20434997
- [Background] Jog MA, Anderson C, Kubicki A, Boucher M, Leaver A, Hellemann G, Iacoboni M, Woods R, Narr K. Transcranial direct current stimulation (tDCS) in depression induces structural plasticity. Sci Rep. 2023 Feb 17;13(1):2841. doi: 10.1038/s41598-023-29792-6. PMID 36801903
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Woodham RD, Rimmer RM, Young AH, Fu CHY. Adjunctive home-based transcranial direct current stimulation treatment for major depression with real-time remote supervision: An open-label, single-arm feasibility study with long term outcomes. J Psychiatr Res. 2022 Sep;153:197-205. doi: 10.1016/j.jpsychires.2022.07.026. Epub 2022 Jul 8. PMID 35839661
- [Background] Woodham RD, Selvaraj S, Lajmi N, Hobday H, Sheehan G, Ghazi-Noori AR, Lagerberg PJ, Rizvi M, Kwon SS, Orhii P, Maislin D, Hernandez L, Machado-Vieira R, Soares JC, Young AH, Fu CHY. Home-based transcranial direct current stimulation treatment for major depressive disorder: a fully remote phase 2 randomized sham-controlled trial. Nat Med. 2025 Jan;31(1):87-95. doi: 10.1038/s41591-024-03305-y. Epub 2024 Oct 21. PMID 39433921
- [Background] Thair H, Holloway AL, Newport R, Smith AD. Transcranial Direct Current Stimulation (tDCS): A Beginner's Guide for Design and Implementation. Front Neurosci. 2017 Nov 22;11:641. doi: 10.3389/fnins.2017.00641. eCollection 2017. PMID 29213226
- [Background] Vogelmann U, Pilloni G, Brunoni AR, Charvet L. How can we develop transcranial direct current stimulation into an effective at-home treatment tool for depression? Expert Rev Med Devices. 2024 Oct;21(10):883-886. doi: 10.1080/17434440.2024.2409767. Epub 2024 Sep 26. No abstract available. PMID 39327744
- [Background] Couture M, Desbeaumes Jodoin V, Bousseau E, Sarshoghi A, Nitsche MA, Blumberger DM, Bolduc C, Weissman CR, Appelbaum LG, Daskalakis ZJ, Poorganji M, Lesperance P, Miron JP. Spaced Transcranial Direct Current Stimulation for Major Depression. Am J Psychiatry. 2025 Mar 1;182(3):276-284. doi: 10.1176/appi.ajp.20240083. Epub 2025 Jan 29. PMID 39876681

DOCUMENTS (1):
  • Informed Consent Form (2025-05-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT07217223/ICF_000.pdf